CLINICAL TRIAL: NCT01484912
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of STA-2 in Patients With Chronic Stable Angina
Brief Title: Phase II Study of STA-2 in Patients With Chronic Stable Angina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinphar Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCCD05014A
Record Dates: First submitted 2007-05-09; First posted 2011-12-02 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Stable Angina
Keywords: Green tea polyphenols; Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — STA 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- STA-2 (Experimental): STA-2 250 mg capsule, each containing 100 mg green tea polyphenols.
  Two capsules t.i.d. (three times daily) for 6 weeks, to be administered in a non-fasting state.
  Interventions: Drug: STA-2
- Placebo (Placebo Comparator): Placebo capsule, containing non-active ingredients.
  Two capsules t.i.d. (three times daily) for 6 weeks, to be administered in a non-fasting state.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STA-2 — After 1 week of screening and washout, patients who met the entry criteria were randomly assigned either to the treatment or control group. The regimen of STA-2 was:
  STA-2 250 mg capsule, each containing 100 mg green tea polyphenols, 2 capsules t.i.d. (three times a day) for 6 weeks, to be administered in a non-fasting state.
  Arms: STA-2
Drug: Placebo — After 1 week of screening and washout, patients who met the entry criteria were randomly assigned either to the treatment or control group. The regimen of Placebo was:
  Placebo 250 mg capsule, 2 capsules t.i.d. (three times a day) for 6 weeks, to be administered in a non-fasting state.
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy, pharmacological activities and safety of STA-2 in the treatment of chronic stable angina.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the efficacy of STA-2 in the management of chronic stable angina. The secondary objectives of this study were to evaluate the safety and pharmacological activities of STA-2 in the management of chronic stable angina. This was a multi-center, double-blind, randomized, parallel-group, placebo-controlled study of STA-2 in the management of chronic stable angina. The study period for each patient was approximately 7 weeks, during which the patient undergone one-week screening and washout period, followed by 6 weeks of treatment. Each patient was required to make a total of 5 visits. Primary Efficacy Endpoint: Change in total exercise time.

After washout, patients who met the inclusion and exclusion criteria were randomly assigned either to the treatment or control group. The respective regimens were:

Treatment group:

STA-2 250 mg capsule, each containing 100 mg green tea polyphenols, 2 capsules ter in die (t.i.d.=three times daily) for 6 weeks, to be administered in a non-fasting state.

Control group:

Placebo 250 mg capsule, 2 capsules t.i.d. (three times daily) for 6 weeks, to be administered in a non-fasting state.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged > 20;
2. Patients who had effort-induced angina which was relieved by rest or nitroglycerin, or who had catheterization-documented coronary artery disease or previous myocardial infarction ≥ 3 months before screening;
3. Patients who manifested positive ETT (exercise tolerance testing) (defined as ST-segment depression ≥ 1 mm compared with at rest, with or without limiting angina) at screening (Day -7);
4. Patients who manifested positive ETT (exercise tolerance testing) (defined as ST-segment depression ≥ 1 mm compared with at rest, with or without limiting angina) on the day of enrollment (Day 0). ETT performance between Day -7 and Day 0 were required not differ by >20% in total exercise time;
5. Female patient who was in the post-menopausal stage or of childbearing potential who:

   * used adequate contraception since last menstruation and no plan for conception during the study;
   * was non-lactating;
   * had negative pregnancy test (urine) within 14 days prior to the study;
6. Able to provide written informed consent.

Exclusion criteria:

1. Patients with pre-excitation, conduction abnormalities, pacemaker rhythm, unstable angina or myocardial infarction within the preceding 3 months;
2. Patients with heart failure (New York Heart Association class III or IV), uncorrected valvular or congenital heart disease, patients who needed digoxin, isosorbide mononitrate, nitroglycerin sustained release preparation, theophylline, class I antiarrhythmic agents, digitalis, or monoamine oxidase inhibitors, as judged by the investigator;
3. Patients with any EKG abnormalities preventing the interpretation of ischemia (complete left bundle branch block);
4. Patients with Chronic Obstructive Pulmonary Disease (COPD) requiring bronchodilators;
5. Patients with hepatic failure (defined as aspartate transaminase (AST) and/or alanine transaminase (ALT) > 3X the upper limit of normal values), and/or renal failure (defined as serum creatinine > 3 mg/dL);
6. Patients with severe gastrointestinal illness as judged by the investigator;
7. Patient with any conditions that interfered the performance of exercise tolerance test as judged by investigator (e.g., knee/ankle arthropathy, Parkinsonism, stroke).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Den Tseng, MD, Ph.D, Principal Investigator — Department of Cardiology National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - Chi Mei Medical Center, Tainan, Tainan
  - National Taiwan University Hospital, Taipei, Taipei
  - Taipei Veterans General Hospital, Taipei, Taipei

REFERENCES:
- [Background] Unno T, Tago M, Suzuki Y, Nozawa A, Sagesaka YM, Kakuda T, Egawa K, Kondo K. Effect of tea catechins on postprandial plasma lipid responses in human subjects. Br J Nutr. 2005 Apr;93(4):543-7. doi: 10.1079/bjn20041379. PMID 15946418
- [Background] Maron DJ, Lu GP, Cai NS, Wu ZG, Li YH, Chen H, Zhu JQ, Jin XJ, Wouters BC, Zhao J. Cholesterol-lowering effect of a theaflavin-enriched green tea extract: a randomized controlled trial. Arch Intern Med. 2003 Jun 23;163(12):1448-53. doi: 10.1001/archinte.163.12.1448. PMID 12824094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Enrolled: May-10-2007 Last Patient Completed: Jun-17-2008
Pre-assignment Details: Patients underwent one-week screening and washout period prior to randomization
Groups:
- STA-2: STA-2 250 mg capsule, each containing 100 mg green tea polyphenols.
  Two capsules three times daily for 6 weeks, to be administered in a non-fasting state.
- Placebo: Placebo capsule, containing non-active ingredients.
  Two capsules three times daily for 6 weeks, to be administered in a non-fasting state.
Period: Overall Study
Arm/Group | STA-2 | Placebo
Started | 39 | 40
Completed | 38 | 39
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STA-2 | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 15 | 16 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 34 | 32 | 66
Region of Enrollment [Number; unit: participants]
  Taiwan | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Exercise Time
Description: Total exercise time was defined as the maximal duration of exercise which was performed by the patient in the setting of exercise tolerance tests (ETT). A 12-lead electrocardiogram (EKG) was used to continuously monitor vital signs. Patients were asked to complete 9-12 minutes of exercise or to exercise until 85% of the maximum predicted heart rate was reached. All exercise tolerance tests used a standard Bruce multistage exercise test protocol.
Time Frame: baseline (visit 2) and week 6 (visit 5)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | STA-2 | Placebo
Number analyzed (Participants) | 38 | 39
seconds | 450.39 (106.7) | 411.15 (118.1)
Statistical Analysis 1: Comparison: STA-2 vs Placebo; T-test was used to compare the change in total exercise time between the treatment groups. The change in total exercise time (△) was defined as the total exercise time at end-point visit minus the total exercise time at baseline. Let △T be the change in total exercise time for treatment group (STA-2) and △C be the change in total exercise time for control group (Placebo). The hypothesis testing for the superiority of STA-2 to Placebo was H0：△T-△C≦0 with H1：△T-△C﹥0; Test type: Non-Inferiority or Equivalence — The superiority testing was conducted one sided with 0.025 significance level. If H0 was rejected one-sided 0.025 significance level, STA-2 was concluded to be statistically superior to Placebo.All hypothesis testing except for the primary efficacy endpoint was conducted two sides at 0.05 significance level and 95% Confidence Interval (C.I.) was adopted if needed; p = 0.025, t-test, 1 sided

2. Secondary Outcome: Changes in Time to 1mm ST-segment Depression During Exercise Tolerance Testing (ETT).
Description: Time to 1 millimeter (mm) ST-segment depression was recorded from Electrocardiogram (EKG) during exercise tolerance testing (ETT). The 1mm ST-segment depression may be seen in typical angina patient. It means the ST segment of EKG wave drops at least 1 mm compared to the beginning of EKG measurement.
Time Frame: baseline (visit 2) through week 6 (visit 5)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | STA-2 | Placebo
Number analyzed (Participants) | 38 | 39
seconds | 396.76 (109) | 341.69 (138.5)
Statistical Analysis 1: Comparison: STA-2 vs Placebo; All hypothesis testing was conducted with T-tests, two sides at 0.05 significance level and 95% Confidence Interval (C.I.) was adopted if needed; Test type: Superiority or Other; p = 0.005, t-test, 2 sided

3. Secondary Outcome: Change in Consumption of Short-acting Nitrates
Description: The consumption of short-acting nitrates from baseline (V2, Day 0) to all visits [V3 (Day 14±2), V4 (Day 28±2), V5 (Day 42±2)]according to patient's diary.
Time Frame: from baseline (visit 2) through week 6 (visit 5)
Reporting Status: Not Posted
Measure: Number (Standard Deviation); unit: participants

4. Secondary Outcome: Change in Rate-pressure Product
Description: Rate-pressure product was defined as the product of heart rate and systolic blood pressure, which was measured both at rest and at peak of exercise.
Time Frame: baseline (visit 2) to week 6 (visit 5)
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: rate

5. Secondary Outcome: Change in Pharmacological Parameters
Description: The level of oxidative stress parameters (isoprostane, homocysteine), homeostasis parameters (PAI-I activity), inflammatory markers (fibrinogen, hsCRP, soluble CD40 ligand) and cardiac enzymes (CPK-MB and LDH), were measured to assess the pharmacological activity of STA-2.
Time Frame: baseline (visit 2) to week 6 (visit 5)
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: stress parameters

6. Secondary Outcome: Consumption of Short-acting Nitrates
Time Frame: The consumption of short-acting nitrates from baseline (V2, Day 0) to all visits [V3 (Day 14±2), V4 (Day 28±2), V5 (Day 42±2)]according to patient's diary.
Population: The data was not available for analysis, because only two patients administered short-acting nitrates
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | STA-2 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | STA-2 | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 1
Other Adverse Events (participants affected / at risk) | 8 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | STA-2 | Placebo
Hospitalization (Surgical and medical procedures) | 0/39 (0) | 1/40 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | STA-2 | Placebo
Palpitations (Cardiac disorders) | 2/39 (2) | 0/40 (0)
chest pain (General disorders) | 2/39 (2) | 0/40 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2/39 (2) | 0/40 (0)
Insomnia (Psychiatric disorders) | 2/39 (2) | 0/40 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No